CLINICAL TRIAL: NCT00586131
Title: Effect of Arterial pH on N-balances of Patients Undergoing Automated Peritoneal Dialysis
Brief Title: Arterial pH and Total Body Nitrogen Balances in APD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 11043
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: End-stage Renal Disease
Keywords: end-stage renal disease; automated peritoneal dialysis; metabolic acidosis; nitrogen balances
MeSH Terms: conditions — Kidney Failure, Chronic; Acidosis | interventions — Ammonium Chloride; Sodium Citrate; Citric Acid

STUDY DESIGN:
Intervention Model Description: Treatment with sodium citrate/citric acid or ammonium chloride chloride in each phase to achieve the desired arterial pH
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low normal pH (arterial pH 7.36-7.38) (Active Comparator): Ammonium chloride or sodium citrate/citrate acid as needed to achieve the target pH
  Interventions: Drug: ammonium chloride or sodium citrate/citric acid
- High Normal pH (arterial pH 7.44-7.46) (Active Comparator): High Normal pH (7.44-7.46) with use of increasing doses of sodium bicarbonate up until the desired pH is achieved
  Interventions: Drug: Sodium citrate/citratic acid

INTERVENTIONS:
Drug: ammonium chloride or sodium citrate/citric acid — Dose dictated by changes in pH
  Arms: Low normal pH (arterial pH 7.36-7.38)
Drug: Sodium citrate/citratic acid — dictated by pH
  Arms: High Normal pH (arterial pH 7.44-7.46)

SUMMARY:
This study will test the hypothesis that by slightly lowering the acidity of blood (or increasing the pH), dialysis patients utilize protein and amino acids more efficiently.

DETAILED DESCRIPTION:
The normal range of pH of the blood (measure of acid-base balance of body) is rather large. It is defined as a range of pH between 7.38 and 7.44. There is evidence to suggest that a high normal arterial pH (7.43-7.45) preserves nutritional status of individuals better than a low normal arterial pH (7.36-7.38). We will test this hypothesis in a small group of stable patients with end-stage renal disease undergoing automated peritoneal dialysis. It needs to be noted that all pH levels to be attained in this study are considered to be normal. The primary outcome measure for the study will be the N-balance. The changes in blood pH will be obtained by medications (ammonium chloride for lower pH and sodium bicarbonate for higher pH).

Study Procedures: A total of eight subjects with end-stage renal disease undergoing automated peritoneal dialysis will be recruited. The initial study procedures will be for purposes of screening individuals for the study. The subjects will perform 24-hour collection of urine and dialysate to assess dialysis dose and a peritoneal equilibration test to evaluate the transport properties of the peritoneum. Only those subjects who receive the minimum dialysis dose and have an average peritoneal transport type will enter the study. During this phase, the subjects will maintain a food diary to evaluate dietary preferences and dietary calorie and protein intake. These data will be used to prepare the diets for the subjects when they are admitted to the GCRC. The next two weeks will be used to evaluate the response of arterial pH to the use of the low alkali solution. If, at the end of two weeks, the arterial pH is not in the desired range, the subjects will require ammonium chloride supplementation to achieve the lower pH. In such subjects, ammonium chloride supplementation will be used for all phases of the study.

Qualifying subjects will be hospitalized in the GCRC for 41 days. The entire period of hospitalization will be divided into two equal phases of 20.5 days each: one will be the low pH phase (low alkali dialysis solution with/without ammonium chloride) and the second will be the high pH phase (high alkali dialysis solution with sodium bicarbonate with/without ammonium chloride). Nitrogen balance will be estimated during the entire period of hospitalization. N-intake is a sum of dietary and medicinal intake, while N-output will be N-losses in dialysate, urine and feces. The N-balance will be the difference between N-intake and N-output. The second outcome measure will be leucine turnover studies. Leucine turnover studies will be performed on days 21 and 41. Leucine turnover studies provide information regarding rates of total body protein synthesis and total body protein degradation as well as rates of leucine oxidation. The study will take 10 hours each - the initial 4 hours will be after an overnight fast and the last six hours will be while being fed. The third outcome measure will be the content of some proteins in a sample of muscle biopsy. Muscle biopsy will be performed on days 21 and 41 after the completion of leucine turnover studies. Finally, nutritional assessment will be performed at the time of patient admission, on day 21 and 41. On days 21 and 41, the nutritional assessment will be performed prior to the start of the leucine turnover studies.

The subjects will be compensated for participation in this study -the amount of compensation will be dependent upon the degree of participation of subjects.

Risk-benefit Assessment: The risks of the study include the risks of performing a muscle biopsy, discomfort associated with the placement of the feeding tube, emotional problems associated with prolonged hospitalization in the GCRC and risks associated with venipuncture. There are no direct benefits to the subjects as a result of their participation in this study. However, if we demonstrate that the higher arterial pH is better at preservation of nutritional status, it may have the potential of decreasing the prevalence and/or severity of protein-energy malnutrition in patients undergoing automated peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from any ethnic/racial group < 65 years.
2. Treatment with CPD for 6 months and current treatment with APD for at least one month.
3. Hemoglobin of at least 11.0 g/dl.
4. Stable dose of erythropoietin treatment for at least the preceding three months.
5. Subjects with normal nutritional status to mild malnutrition:

   1. Serum albumin > 3.3 g/dl
   2. Relative body weight of 90-120% of the NHANES II median body weight for a given height, age range, gender and frame size.
   3. A normalized protein equivalent of total nitrogen appearance (nPNA) > 0.80 g/kg actual body weight/day at the time of screening.
6. D/P Cr between 0.48 and 0.81 on the PET performed at the time of the screen.
7. Total (renal + peritoneal) weekly Kt/V urea > 1.70 and creatinine clearance > 50 L/wk/1.73 m2.
8. No evidence of primary or secondary (viz., ischemic, neuropathic) myopathy

Exclusion Criteria:

1. History of active cancer other than basal cell carcinoma.
2. Symptomatic severe ischemic heart disease, uncontrolled severe dysrhythmias, uncontrolled congestive heart failure, poorly controlled hypertension, severe musculoskeletal disease, arthritis or amputation of the lower extremities.
3. Insulin requiring diabetes mellitus.
4. Patients who received L-carnitine or anabolic hormones (other than erythropoietin) within the previous 6 months.
5. Use of CaCO3 as phosphate binder.
6. Severe lung or liver disease, uncontrolled asthma, active vasculitis.
7. Severe chronic infection or any other acute or chronic inflammatory or catabolic illnesses (e.g., active tuberculosis, AIDS, osteomyelitis).
8. Psychosis, inability to give informed consent, evidence that patient will not comply with study protocol.
9. Alcohol or other recreational drug abuse.
10. Pregnancy (rare in CPD patients).
11. Patients who are physically and/or psychologically incapable of undergoing the protocol.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
N-balances | 20 days
  Total body nitrogen balance defined as difference between nitrogen intake and nitrogen appearance in urine, stool, and dialysate

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mehrotra, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

REFERENCES:
- [Derived] Mehrotra R, Bross R, Wang H, Appell M, Tso L, Kopple JD. Effect of high-normal compared with low-normal arterial pH on protein balances in automated peritoneal dialysis patients. Am J Clin Nutr. 2009 Dec;90(6):1532-40. doi: 10.3945/ajcn.2009.28285. Epub 2009 Oct 21. PMID 19846545